CLINICAL TRIAL: NCT06248073
Title: Comparing the Effectiveness of Online Self-management Program and On-site Task-related Training for People With Early Stage Parkinson's Disease on Activity Participation and Quality of Life
Brief Title: Effectiveness of Online Program and Task-related Training for Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Kuan-yi Li, Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202202160B0C601
Record Dates: First submitted 2024-01-07; First posted 2024-02-08 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease; Occupational Therapy; Telerehabilitation; Activities of Daily Living
Keywords: Telerehabilitation; early intervention; patient-reported outcome assessment; self-perception
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- on-line self-management group (Experimental): The investigators plan to conduct 12 sessions of intervention, one hour per session, 2 sessions per week, for a total of 6 weeks. Participants will receive interventions in their home via online meetings with a certified occupational therapist. The training will be related to functional tasks in daily life. In addition, the investigators will guide participants to use self-management skills in their daily routines. Participants will receive booklets to conduct their self-practice and exercise for 30 minutes per session, two sessions per week, for a total of 6 weeks.
  Interventions: Behavioral: on-line self-management training
- on-site task-related group (Experimental): The investigators plan to conduct 12 sessions of intervention, one hour per session, 2 sessions per week, for a total of 6 weeks. Participants will receive interventions at Chang Gung Memorial Hospital. A certified occupational therapist will conduct the interventions. The training will include motor function of upper extremities, balance training and functional tasks. The level of difficulty of the tasks will be adjusted based on the participants' abilities.
  Interventions: Behavioral: onsite task-related training
- control group (No Intervention): To compare the two experimental groups in the context of early Parkinson's disease, the control group will not receive any additional intervention and will continue their regular daily activities without changes.

INTERVENTIONS:
Behavioral: on-line self-management training — To encourage adherence to the home program among early-stage Parkinson's disease participants, the investigators have developed various self-management topics, including medication adherence and exercise benefits. The home program is categorized into two dimensions: daily function and exercise. The investigators will provides participants with detailed guidelines to ensure safe execution of the program independently.
  Arms: on-line self-management group
Behavioral: onsite task-related training — Participants will receive interventions at Chang Gung Memorial Hospital. A certified occupational therapist will conduct the interventions. These sessions will involve functional tasks tailored to each participant's skill level, with two to four varied tasks per session. Additionally, participants will be given booklets to guide them in self-managing similar exercises at home, mirroring the home program of the self-management group.
  Arms: on-site task-related group

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of online self-management program and on-site task-related training for people with early stage Parkinson's disease.

people with early stage of Parkinson's disease (age range: 45-70 years) will be randomly assigned into the following three groups: control group, online self-management program group and on-site task-related training group.The control group will receive no treatment during the experimental period. For the other two groups, participants will receive the intervention twice a week, one hour per session and 12 sessions in total.

The main questions it aims to answer are:

1. the potential impact of motor and non-motor symptoms on activity participation and quality of life for people with early stage of Parkinson's disease (PD).
2. compare and examine the the effectiveness of online self-management program and on-site task-related training for people with early stage Parkinson's disease on activity participation and quality of life.

DETAILED DESCRIPTION:
This study aims to answer two major research questions. First, the investigators will investigate the potential impact of motor and non-motor symptoms on activity participation and quality of life for people with early-stage Parkinson's disease (PD). Second, the investigators will compare and examine the effectiveness of online self-management programs and on-site task-related training for people with early-stage Parkinson's disease on activity participation and quality of life.

Introduction: Previous studies have indicated that hand function impairment may be one of the early motor symptoms and precursor markers of Parkinson's disease. Compared to only receiving drug treatment, additional interventions such as exercise training, environmental adjustments, cognitive behavior and self-management can effectively improve the execution of daily activities and improve the quality of life of patients.

Method: The investigators plan to recruit 100 participants within three years and randomly assign them to one of the following three groups: control group, online self-management program group, and on-site task-related training group.

Participants: People with early-stage Parkinson's disease (age range: 45-70 years).

Procedure: The control group will receive no treatment during the experimental period. For the other two groups, participants will receive the intervention twice a week, one hour per session, and 12 sessions in total. The online self-management program will be an individualized self-management program provided remotely by certified occupational therapists. The on-site task-related training program will include balance and exercise, hand function, and functional task training.

Outcome measures: The assessment will be performed before intervention, after the completion of intervention, and 6 months after the post-test. Prior to the experiment, the investigatorswill conduct a pretest. Then, the investigators will conduct a post-test (after intervention) to ensure the short-term effects.

Follow-up: After six months of completing the post-test, the cases will undergo a second post-test to understand the long-term effects.

Statistical analysis: This study will use two-way repeated measured ANOVA design.The independent variables consist of two factors: the first is the between-group factor, which is the intervention method (control group vs.online self-management program group vs. physical task-related training group); the second is the within-group factor, which is time (pretest vs. first post-test vs. second post-test (follow-up).

ELIGIBILITY:
Inclusion criteria:

1. Willingness to sign the informed consent form.
2. Age between 45 and 70 years, with mild idiopathic Parkinson's disease and Hoehn and Yahr stage 1-2.
3. No cognitive impairment.
4. No severe depression that could affect the motivation to participate in the study.
5. No history of shoulder dislocation or fracture that could affect body proprioception.
6. No diseases that could affect the ability to reach for objects, such as stroke.
7. No diseases that could affect peripheral sensation, such as diabetes.
8. No severe tremors; patients whose hands, when relaxed and placed on the apparatus, still exhibit significant tremor interfering with the experiment will not be included.
9. Able to follow instructions and complete the assessment process.
10. Have not received physical or occupational therapy in the past year.

Exclusion criteria:

1. Other central nervous system diseases, such as stroke.
2. Have major surgery on the head or upper limbs.
3. Inability to perform the reaching task while sitting.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Purdue Pegboard Test | Baseline (before intervention), week 6 (after intervention), follow-up (6 months after intervention)
  The change from baseline in dexterity will be measured by the number of pegs participants can put into the holes as quickly as possible. The higher the score, the better the hand dexterity. The test consists of four tasks: inserting pegs with the right hand, inserting pegs with the left hand, inserting pegs with both hands, and assembling pegs with both hands. The time taken to complete the test will be recorded.
Box and Block test | Baseline (before intervention), week 6 (after intervention), follow-up (6 months after intervention)
  The change from baseline in dexterity will be measured by the number of blocks participants can put to another box as quickly as possible. Box and Block test is a commonly used tool in occupational therapy to assess hand dexterity. The patient is seated and the experimenter sits opposite the patient to confirm the testing process. The patient is asked to perform the test with their dominant hand, picking up one block at a time and crossing the partition with the block, placing it in the empty space on the other side. The faster the better. Before the formal test, the patient is given 15 seconds of practice time. The formal test lasts for 1 minute.
Proprioceptive sensitivity Assessment | Baseline (before intervention), week 6 (after intervention), follow-up (6 months after intervention)
  The examiner will use a customized apparatus from the Sensorimotor Control Laboratory at the University of Minnesota to assess position sense motion sense acuity. Participants will be tested on the same-side position matching test and the psychophysical discrimination threshold test. The examiner moves the examinee's testing hand from the starting position to the testing position and then moves the examinee's wrist back to the starting position.
  The instrument will use an adaptive algorithm to determine whether to give a simpler or more difficult displacement for the next trial based on whether the examinee's answer is correct or not. A total of about 20 tests are required, and the test time is about 10-15 minutes. The instrument will record the position matching error.
Nottingham Extended Activities of Daily Living Scale (NEADL) | Baseline (before intervention), week 6 (after intervention), follow-up (6 months after intervention)
  This assessment tool is used to measure an individual's capacity for instrumental activities of daily living. Based on the classification of the International Classification of Functioning, Disability, and Health (ICF model), the assessment pertains to the level of activities and participation. It includes a total of 22 items, all of which are activities performed in daily life. Participants are asked to respond based on their actual performance or involvement in these activities over the past few weeks. Each item has four response options for the participant to self-report: can complete independently, can complete independently but with some difficulty, requires assistance from others to complete, and did not perform this activity. Each item is scored on a scale of 0-3, with a total score of 66. The higher the score, the better the patient's ability to perform daily activities of living.
Parkinson's Disease Questionnaire (PDQ-39) | Baseline (before intervention), week 6 (after intervention), follow-up (6 months after intervention)
  This self-administered questionnaire consists of 39 questions assessing the quality of life of individuals with Parkinson's disease across eight dimensions, including mobility, activities of daily living, emotional wellbeing, stigma, cognition, social support, communication, and bodily discomfort. The questions ask participants to rate the difficulty they experienced in various activities during the past month of living with Parkinson's disease. There are five response options for each question: Not at all, Occasionally, Sometimes, Often, and Always or cannot do at all, scored from 0 to 4, respectively. A higher score indicates greater difficulty experienced by the participant.

SECONDARY OUTCOMES:
Time up and go test (TUG) | Baseline (before intervention), week 6 (after intervention), follow-up (6 months after intervention)
  The change from baseline in mobility will be measured by the time taken as recorded. Before the test, the examinee sits steadily, readying for the test. Upon the examiner's cue, they stand from the chair and walk three meters, then turn, and sit back down. This duration is timed with a stopwatch by the examiner. To ensure accuracy, the test is repeated three times, averaging the times. The Timed Up and Go test serves as a swift, practical method for assessing functional mobility and pinpointing those at heightened fall risk or needing additional balance or gait training.
Grip Strength measure | Baseline (before intervention), week 6 (after intervention), follow-up (6 months after intervention)
  The change from baseline in grip strength will be measured by the mean values to the norm according to participant's age and gender. The participant should sit with their upper arms naturally hanging down and their elbows bent at a 90-degree angle. Then, the participant should measure their grip strength three time, and the average of the three measurements should be analyzed.
Pinch Strength measure | Baseline (before intervention), week 6 (after intervention), follow-up (6 months after intervention)
  The change from baseline in pinch grip will be measured by the mean values to the norm according to participant's age and gender. The participant should sit with their upper arms naturally hanging down and their elbows bent at a 90-degree angle. Then, the participant should measure their lateral /key pinch and palmar /three-jaw chuck pinch strength three times each, and the average of the three measurements for each method should be analyzed.
Hand length measure | Baseline (before intervention)
  Hand length is measured at baseline to provide information for adjusting the value of strength during statistical analysis. To measure the length of the hand, ask the participant to place their palm flat and facing up, and then measure the distance from the tip of the middle finger to the wrist crease.
The University of Pennsylvania Smell Inventory Test (UPSIT) | Baseline (before intervention), week 6 (after intervention), follow-up (6 months after intervention)
  Olfactory function can be tested using standardized quantitative assessment tools. Commonly used in research are the University of Pennsylvania Smell Identification Test (UPSIT) and the smell threshold test. The method of testing smell identification primarily involves forty different scents. Test participants are required to smell the odors presented on each page of the test booklet and choose the correct answer from four options. Each item is scored one point, with a total possible score of forty. A higher score indicates better smell identification ability.
Montreal Cognitive Assessment (MoCA) | Baseline (before intervention)
  This measurement is used to assess the cognitive function of participants and can effectively distinguish mild cognitive impairments. Initially developed for the diagnosis of dementia, it has since been widely used. The test takes about 10 minutes and measures seven cognitive domains, including visual-spatial/executive functions, naming, verbal memory registration and learning, attention, language, delayed memory, abstract thinking, and orientation. Each domain is scored differently, with the total score ranging from 0 to 30 points. Additionally, considering the impact of educational level, one extra point is added for individuals with less than 12 years of education. Lower scores indicate more severe cognitive impairment.
International Physical Activity Questionnaire (IPAQ) | Baseline (before intervention), week 6 (after intervention), follow-up (6 months after intervention)
  The change from baseline in physical activity will be measured by IPAQ scores. Taiwan version has been testified validity and reliability. This questionnaire including four domains: Job, Transportation, Housework, Leisure. Duration and frequency of physical activity in the last 7 days will be measured.
The Pittsburgh Sleep Quality Index (PSQI) | Baseline (before intervention), week 6 (after intervention), follow-up (6 months after intervention)
  The change from baseline in sleep quality will be measured by PSQI scores. It is a self-rated questionnaire that assesses sleep quality over the past month. It consists of ten questions and covers various aspects of sleep such as sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. The questionnaire has 19 individual items, 7 component scores, and each item is scored on a scale of 0 to 3. Higher scores indicate worse sleep quality.
WHOQOL-bref Taiwan version | Baseline (before intervention), week 6 (after intervention), follow-up (6 months after intervention)
  The change from baseline in quality of life will be measured by WHOQOL-bref scores.The questionnaire is simplified from the original six domains to four domains. This is a self-reported questionnaire that assesses quality of life based on personal feelings and subjective experiences in the past two weeks. It consists of 28 questions, each scored using a Likert scale with five points. The questionnaire covers four major domains: physical, psychological, social relationships, and environmental interactions. A higher score indicates a better quality of life.
Multidimensional Fatigue Inventory (MFI) | Baseline (before intervention), week 6 (after intervention), follow-up ( 6 months after intervention)
  The change from baseline in degree of fatigue will be measured by MFI total score. MFI is a self-administered questionnaire that asks the individual to recall their fatigue levels over the past two weeks. The questionnaire consists of 20 questions, including five dimensions of fatigue: general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue. Each question is scored using a Likert scale ranging from 1 (strongly agree) to 5 (strongly disagree).
Home activity log | Within the intervention (6 weeks)
  A customized diary format is utilized to aid participants in executing participants' self-management plans. It will be used within 6 weeks (within the intervention). The participants have to record their exercises each time (at least twice a week). The format encompasses logging dates, frequency, and duration of activities performed at home, along with any challenges or difficulties faced. These details are subsequently reviewed with the therapist in follow-up sessions.
General Self-Efficacy Scale (GSE) | Baseline (before intervention), week 6 (after intervention), follow-up ( 6 months after intervention)
  The change from baseline in self-efficacy will be measured by GSE total score. The purpose of this test is to understand the individual's self-efficacy. The questionnaire consists of 10 items that assess the individual's feelings, thoughts, and actions. Each item is scored on a 4-point scale, with 1 indicating "completely incorrect," 2 indicating "somewhat correct," 3 indicating "mostly correct," and 4 indicating "completely correct." The final score is calculated by summing up the scores of all items. A higher score indicates better self-efficacy.
The unified Parkinson's disease rating scale (UPDRS) | Baseline (before intervention), week 6 (after intervention), follow-up (6 months after intervention)
  The change from baseline in motor function will be measured by the motor subscore and disease severity will be measured by total scores of UPDRS. UPDRS is the most widely used clinical rating scale for Parkinson's disease.This scale is divided into four sections: The first covers mentation, behavior, and mood; the second assesses daily living activities; the third focuses on motor examination; and the fourth evaluates treatment complications. The lowest score is 0, indicating an absence of signs and symptoms of Parkinson's disease.

OTHER OUTCOMES:
Mini-Mental Status Examination (MMSE) | Screening-before intervention (one of the inclusive criteria)
  To ensure participants do not have dementia or other cognitive impairments. The scale consists of 20 questions and 30 items, including orientation, memory, attention and calculation, recall, and language ability. Each correct answer is scored 1 point, and incorrect or unanswerable questions are scored 0 points. The total score ranges from 0 to 30 points. Lower score indicates more severe cognitive impairment.
Beck depression scale | Screening-before intervention (one of the inclusive criteria)
  The objective is to confirm that study participants do not suffer from severe depression. Should severe depression be detected in a potential participant, they will be excluded from recruitment. The scale consists of 21 questions and 30 items, with a total score of 63 points. A score of 14-19 indicates mild depression, 20-28 indicates moderate depression, and 29 or higher indicates severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-yi Li, PhD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital, Linkou District, Taiwan

IPD SHARING:
Plan to Share IPD: No